CLINICAL TRIAL: NCT07381686
Title: High-Flow Nasal Cannula Versus Noninvasive Ventilation After Extubation in Patients With COPD and Mild Hypercapnic Respiratory Failure: A Prospective, Randomized Comparative Study
Brief Title: High-Flow Nasal Cannula Versus Noninvasive Ventilation After Extubation in Patients With COPD and Mild Hypercapnic Respiratory Failure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Montaser Gamal Ahmed, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFNC vs NIV in COPD weaning
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: COPD
Keywords: NIV,HFNC
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIV group (Experimental): using Non-Invasive Ventilation (NIV) as the intervention device, a BiPAP machine will be used with an oronasal mask, adjusting inspiratory and expiratory pressures based on patient tolerance and ABG results.
  Interventions: Device: Non-Invasive Ventilation (NIV)
- HFNC group (Experimental): using High-Flow Nasal Cannula (HFNC) as intervention device, Patients assigned to the HFNC arm will receive oxygen through a high-flow nasal cannula connected to a heated humidifier, with flow rates titrated up to 60 L/min and FiO₂ adjusted to maintain target oxygen saturation (88-92%).
  Interventions: Device: High-Flow Nasal Cannula (HFNC)

INTERVENTIONS:
Device: Non-Invasive Ventilation (NIV) — In the NIV group, a BiPAP machine will be used with an oronasal mask, adjusting inspiratory and expiratory pressures based on patient tolerance and ABG results.
  Arms: NIV group
Device: High-Flow Nasal Cannula (HFNC) — Patients assigned to the HFNC arm will receive oxygen through a high-flow nasal cannula connected to a heated humidifier, with flow rates titrated up to 60 L/min and FiO₂ adjusted to maintain target oxygen saturation (88-92%).
  Arms: HFNC group

SUMMARY:
Acute exacerbations of chronic obstructive pulmonary disease (AECOPD) represent a leading cause of hospital admissions and respiratory intensive care unit (RICU) stays worldwide. After invasive mechanical ventilation, many COPD patients experience difficulty in the weaning process, with a high hazard of extubation failure due to persistent hypercapnia and weakened respiratory muscle function (1). Extubation failure is allied with increased morbidity, prolonged ICU stay, and higher mortality (2). Thus, effective post-extubation respiratory support strategies are central for improving outcomes in this susceptible group.

Conventionally, noninvasive ventilation (NIV) has been the standard of care after extubation in COPD patients with mild to moderate hypercapnic respiratory failure, as it decreases work of breathing, improves gas exchange, and lowers reintubation rates (4). Though, NIV can be poorly tolerated due to mask-related discomfort, skin breakdown, claustrophobia, and patient-ventilator asynchrony (4).These limits often lead to suboptimal adherence and may compromise its efficacy in practice.

High-flow nasal cannula (HFNC) oxygen therapy has arisen as another, offering heated and humidified oxygen at high flows, which provides low-level positive airway pressure, washes out nasopharyngeal dead space, and improves patient comfort (5). Recent trials suggest that HFNC may be non-inferior to NIV in preventing post-extubation respiratory failure in high-risk populations (6). Yet, data specifically addressing COPD patients with mild hypercapnic respiratory failure remain inadequate, and no agreement exists regarding the optimal strategy in this subgroup. Thus, a direct comparative study between HFNC and NIV in this context is reasonable to guide clinical practice (7).

DETAILED DESCRIPTION:
Acute exacerbations of chronic obstructive pulmonary disease (AECOPD) represent a leading cause of hospital admissions and respiratory intensive care unit (RICU) stays worldwide. After invasive mechanical ventilation, many COPD patients experience difficulty in the weaning process, with a high hazard of extubation failure due to persistent hypercapnia and weakened respiratory muscle function (1). Extubation failure is allied with increased morbidity, prolonged ICU stay, and higher mortality (2). Thus, effective post-extubation respiratory support strategies are central for improving outcomes in this susceptible group.

Conventionally, noninvasive ventilation (NIV) has been the standard of care after extubation in COPD patients with mild to moderate hypercapnic respiratory failure, as it decreases work of breathing, improves gas exchange, and lowers reintubation rates (4). Though, NIV can be poorly tolerated due to mask-related discomfort, skin breakdown, claustrophobia, and patient-ventilator asynchrony (4).These limits often lead to suboptimal adherence and may compromise its efficacy in practice.

High-flow nasal cannula (HFNC) oxygen therapy has arisen as another, offering heated and humidified oxygen at high flows, which provides low-level positive airway pressure, washes out nasopharyngeal dead space, and improves patient comfort (5). Recent trials suggest that HFNC may be non-inferior to NIV in preventing post-extubation respiratory failure in high-risk populations (6). Yet, data specifically addressing COPD patients with mild hypercapnic respiratory failure remain inadequate, and no agreement exists regarding the optimal strategy in this subgroup. Thus, a direct comparative study between HFNC and NIV in this context is reasonable to guide clinical practice (7).

ELIGIBILITY:
1. Age ≥ 18 years.
2. Established COPD diagnosis (clinical history + prior spirometry confirming persistent airflow limitation, if available).
3. Recently extubated after invasive mechanical ventilation for an acute COPD exacerbation.
4. Mild hypercapnic respiratory failure post-extubation, defined as: PaCO₂ 45-60 mmHg (or ≥10 mmHg above known baseline) and pH ≥ 7.30, and Respiratory rate ≥ 20/min or increased work of breathing.
5. Hemodynamic stability: MAP ≥ 65 mmHg without escalating vasopressors.
6. Adequate airway protection: GCS ≥ 13, no active vomiting, manageable secretions.
7. Oxygenation compatible with noninvasive support (e.g., SpO₂ ≥ 88-92% achievable with FiO₂ ≤ 0.6 during screening).
8. Ability to give informed consent (patient or legal surrogate).

Exclusion criteria:

1. Severe acidosis or severe hypercapnia: pH < 7.30 or PaCO₂ > 60 mmHg requiring immediate escalation.
2. Impending respiratory arrest or immediate need for re-intubation (severe hypoxemia, refractory distress, profound altered mental status).
3. Severe hypoxemia not compatible with trial modalities (e.g., need for FiO₂ > 0.8 or PEEP > 10 cmH₂O to keep SpO₂ ≥ 88%).
4. Hemodynamic instability: shock with rapidly escalating vasopressors, malignant arrhythmia, or active myocardial ischemia.
5. Severe encephalopathy (GCS < 13) or inability to protect airway.
6. Massive hemoptysis, active upper GIT bleeding, or untreated pneumothorax.
7. Post-extubation laryngeal edema/stridor requiring immediate re-intubation.
8. Absolute/relative contraindications to NIV (mask-based): facial trauma/burns, recent facial/upper airway or gastric surgery, fixed upper airway obstruction, uncontrolled vomiting, severe agitation or mask intolerance.
9. Contraindications to HFNC judged by the treating team (rare; e.g., complete nasal obstruction).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Extubation failure (need for reintubation within 72 hours). | within 72 hours.

CONTACTS AND LOCATIONS:
Overall Officials: montaser gamal ahmed, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, أسيوط - Asyut Governorate, Egypt